CLINICAL TRIAL: NCT05456893
Title: A Multicentre Prospective Longitudinal Observational Study to Evaluate Biomarkers in Moderate to Severe Ulcerative Colitis (UC) Patients Treated With Different Targeted Therapies
Brief Title: A Study to Evaluate Biomarkers in Moderate to Severe Ulcerative Colitis (UC) Patients Treated With Different Targeted Therapies
Acronym: ImmUniverse
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Laurent PEYRIN-BIROULET, Principal Investigator (France), Central Hospital, Nancy, France
Other Study IDs: 021-A01092-39
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
Keywords: Ulcerative Colitis; Immune-Mediated Inflammatory Diseases; Biomarkers
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling (RNA and DNA profiling, PBMC isolation, Immunophenotyping, serum and plasma markers) Endoscopic biopsy sampling : Healthy and lesion area (DMSO) Stool sampling (RNA later)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UC patients: All patients with an established ulcerative colitis
  Interventions: Procedure: Procedure: endoscopic biopsy; Procedure: Blood sampling; Procedure: stool sampling

INTERVENTIONS:
Procedure: Procedure: endoscopic biopsy — Per-endoscopic biopsies
Procedure: Blood sampling — Blood sampling
Procedure: stool sampling — stool sampling

SUMMARY:
UC is a chronic, idiopathic form of intestinal inflammatory disease (IBD) that affects the colon, most commonly afflicting adults aged 30-40 years and resulting in disability and lower quality of life (1). It is characterized by relapsing and remitting mucosal inflammation, starting in the rectum and extending to proximal segments of the colon. Although biologic therapies have provided clinical benefits to patients, these goals are still poorly met, due to the limited knowledge of the underlying mechanisms of immunopathology and the lack of predictive biomarkers that would allow proper patient stratification.

The hypothesis of this study is that by identifying new biomarkers in blood, stool and tissue that (i) predict response (or non-response) to therapy prior to the start of treatment and (ii) predict response to therapy in the early phase of treatment will allow to find the right treatment for the right patient (personalized medicine).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 years of age (at the time of signing the ICF)
* Established diagnosis of ulcerative colitis with a minimum disease duration of 3 months
* Moderate to severe active UC defined by Mayo Score ≥ 6
* Moderate to severe active UC defined by endoscopy score of ≥2
* Indication to start any biological or small molecule agent (anti-TNF, anti- IL12/23, anti-integrin and JAK-inhibitors)
* In case of treatment with corticosteroid: stable dose for at least 3 weeks prior to baseline, dosage ≤ 20 mg prednisone
* Indication for an endoscopy for the assessment of disease activity as for standards of care and current guidelines
* Able to comply with the study procedures
* Person affiliated to or beneficiary of a social security plan
* Person informed about study organization and able to sign informed consent form

Exclusion Criteria:

* Diagnosis of indeterminate colitis, microscopic colitis, ischaemic colitis, infectious colitis, radiation colitis
* Absolute contraindications to endoscopy procedures or complication during previous endoscopy
* Bleeding disorders
* Indication for surgery for UC
* Rectal topical therapy (enemas or suppositories) ≤ 2 weeks prior to baseline
* Treatment with > 20 mg prednisone within 3 weeks prior to baseline
* Anaemia (haemoglobin < 10 g/dl) at baseline
* Any circumstances which could contradict a study participation and lead the Investigator to assess the patient as unsuitable for study participation for any other reason
* Person referred in articles L.1121-5, L. 1121-7 and L.1121-8 of the Public Health Code:

  * Pregnant, parturient or breastfeeding woman
  * Minor person (non-emancipated)
  * Adult person under legal protection (any form of public guardianship)
  * Adult person incapable of giving consent and not under legal protection
* Person deprived of liberty for judicial or administrative decision, person under psychiatric care as referred in articles L. 3212-1 and L. 3213-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe active UC with an indication to start a biologic treatment.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2027-09-09 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects who achieve clinical response at week 14. | The percentage of subjects who achieve clinical response at week 14
  Clinical response will be defined as overall Mayo score of 2 or smaller with Mayo endoscopy score (Mayo ES) of 0 or 1 (without friability), and bleeding subscore of 0.
  The Clinical Response will be categorized in four subcategories:
  * Super responder: meets criteria of clinical response
  * Responder: Mayo Score: reduction of 50%/ improvement of ≥ 3 from baseline, but does not meet criteria of remission; endoscopic Mayo: does not meet criteria of clinical response, but shows reduction of Mayo ES
  * Partial responder: Mayo Score: reduction of up to 30%, endoscopic Mayo: no formal improvement by Mayo ES but in overall assessment by the physician slight improvement.
  * Non-responder: reduction of less than 30% and in endoscopy no improvement in the overall assessment
The percentage of subjects who achieve deep clinical remission at week 14. | The percentage of subjects who achieve deep clinical remission at week 14
  Deep clinical remission will be defined as partial Mayo Score 0-1 with stool frequency (SF) ≤1 and rectal bleeding (RB) = 0.
The percentage of subjects who achieve deep clinical remission at week 26. | The percentage of subjects who achieve deep clinical remission at week 26.
  Deep clinical remission will be defined as partial Mayo Score 0-1 with stool frequency (SF) ≤1 and rectal bleeding (RB) = 0.
The percentage of subjects who achieve deep clinical remission at week 52. | The percentage of subjects who achieve deep clinical remission at week 52.
  Deep clinical remission will be defined as partial Mayo Score 0-1 with stool frequency (SF) ≤1 and rectal bleeding (RB) = 0.
The percentage of subjects who achieve mucosal healing at week 14. | The percentage of subjects who achieve mucosal healing at week 14.
  Mucosal healing will be defined as Mayo endoscopic score = 0; Nancy histology index: ulceration: 0, neutrophils: 0, chronic infiltrate: 0 or 1.
The percentage of subjects who achieve mucosal healing at week 52. | The percentage of subjects who achieve mucosal healing at week 52.
  Mucosal healing will be defined as Mayo endoscopic score = 0; Nancy histology index: ulceration: 0, neutrophils: 0, chronic infiltrate: 0 or 1.
The percentage of subjects who achieve symptomatic remission at week 14. | The percentage of subjects who achieve symptomatic remission at week 14.
  Symptomatic remission will be defined as reported by patient on PRO 2 (SF= 0-1 and RB= 0).
The percentage of subjects who achieve symptomatic remission at week 26. | The percentage of subjects who achieve symptomatic remission at week 26.
  Symptomatic remission will be defined as reported by patient on PRO 2 (SF= 0-1 and RB= 0).
The percentage of subjects who achieve symptomatic remission at week 52. | The percentage of subjects who achieve symptomatic remission at week 52.
  Symptomatic remission will be defined as reported by patient on PRO 2 (SF= 0-1 and RB= 0).

SECONDARY OUTCOMES:
The percentage of subjects without any disease progression (e.g. flares) at week 14. | The percentage of subjects without any disease progression (e.g. flares) at week 14.
  The percentage of subjects without any disease progression (e.g. flares) at week 14.
The percentage of subjects without any disease progression (e.g. flares) at week 26. | The percentage of subjects without any disease progression (e.g. flares) at week 26.
  The percentage of subjects without any disease progression (e.g. flares) at week 26.
The percentage of subjects without any disease progression (e.g. flares) at week 52. | The percentage of subjects without any disease progression (e.g. flares) at week 52.
  The percentage of subjects without any disease progression (e.g. flares) at week 52.
The percentage of subjects who show an improvement on patient reported outcomes at week 14. | The percentage of subjects who show an improvement on patient reported outcomes at week 14.
  Patient reported outcomes include: PRO 2 (stool frequency (SF) and rectal bleeding (RB)), FACIT-F (level of fatigue), PROMIS Depression (level of depression), SF-36 (level of quality of life), Euro-QoL-5D (level of quality of life).
The percentage of subjects who show an improvement on patient reported outcomes at week 26. | The percentage of subjects who show an improvement on patient reported outcomes at week 26.
  Patient reported outcomes include: PRO 2 (stool frequency (SF) and rectal bleeding (RB)), FACIT-F (level of fatigue), PROMIS Depression (level of depression), SF-36 (level of quality of life), Euro-QoL-5D (level of quality of life).
The percentage of subjects who show an improvement on patient reported outcomes at week 52. | The percentage of subjects who show an improvement on patient reported outcomes at week 52.
  Patient reported outcomes include: PRO 2 (stool frequency (SF) and rectal bleeding (RB)), FACIT-F (level of fatigue), PROMIS Depression (level of depression), SF-36 (level of quality of life), Euro-QoL-5D (level of quality of life).
The percentage of subjects without the following complications until week 52 : | week 52
  The percentage of subjects without the following complications until week 52:
  * hospitalizations due to UC
  * treatment intensification including introduction of toxic long-term therapies (i.e. systemic glucocorticoids)
  * new stenosis
  * new fistula
  * new development of primary sclerosing cholangitis (PSC)
  * infections
  * intestinal surgery
The percentage of subjects without long-term complications until week 104. | The percentage of subjects without long-term complications until week 104.
  The percentage of subjects without long-term complications until week 104.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan MD SCHREIBER, PhD, Study Director — Christian Albrechts Universität
Locations (1):
- Central Hospital, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No